CLINICAL TRIAL: NCT05187065
Title: The Effect of Mobile-based Education and Exercise Program Given to Patients With Total Knee Replacement Surgery on Anxiety, Kinesiophobia, and Physical Function
Brief Title: The Effect of Mobile-based Education and Exercise Program Given to Patients With Total Knee Replacement Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alkay Kara (Other)
Responsible Party: Sponsor-Investigator, Alkay Kara, Principal Investigator, Giresun University
Organization: Giresun University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: A-KARA-001
Record Dates: First submitted 2021-12-24; First posted 2022-01-11 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Replacement, Knee
Keywords: Mobile based application; Progressive relaxation exercise; Knee exercise; Kinesiophobia; Patient Education; Physical Function; Sleep Quality; Pain; Nursing
MeSH Terms: conditions — Kinesiophobia; Sleep Initiation and Maintenance Disorders; Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile-based education and exercise program (Experimental): Mobile-based education and progressive relaxation and knee exercise program will be applied to the patients in the experimental group.
  Interventions: Other: The mobile-based education and exercise program
- Standard of care (No Intervention): Mobile-based education and progressive relaxation and knee exercise program will not be applied to the patients in the control group, and the clinical routine will be maintained.

INTERVENTIONS:
Other: The mobile-based education and exercise program — Starting from the preoperative period, mobile-based patient education, progressive relaxation exercise and knee exercise program will be applied to the patient as a whole. Mobile-based education will include pre-operative and discharge education. The patient will be given a progressive relaxation exercise with the support of the mobile application and the exercises included in the knee exercise program that should be done after the surgery will be shown. Progressive relaxation exercises will be applied twice a day in the afternoon and evening. Postoperative knee exercises will be performed 3 to 5 times a day, depending on the type of exercise. These exercises will be continued regularly for up to 4 weeks after discharge.
  Arms: Mobile-based education and exercise program

SUMMARY:
Total knee replacement (TDP) surgery is recognized as an effective surgical option for patients who develop moderate to severe osteoarthritis of the knee. Before, during and after TDP surgery, patients experience physical, psychological and social problems. After TDP surgery, patients may experience problems such as dependency and sleep problems in their daily living activities. Patients who have sleep problems, who cannot rest enough, become tired and experience anxiety as a result. It has been stated that the education given to the patients in the preoperative period reduces anxiety and analgesic needs and increases satisfaction. Progressive relaxation exercises in patients It has been shown to be effective in reducing symptoms such as anxiety, pain and fatigue. With the widespread use of mobile technologies, a rapid development is observed in mobile health applications and it is thought that its use in the field of health will provide great benefits to nursing services. This study is of the randomized controlled experimental type. During the application process, a mobile-based training and exercise program will be applied to the patients in the experimental group. As the education content, information about pre- and post-operative information and video-supported training content that will guide the patients with voice commands about the exercises that the patients will do before the surgery will be included in the mobile application. With the implementation of this program, continuity will be ensured by meeting the information needs of the patients before and after the surgery, and by performing progressive relaxation and knee exercises correctly and regularly. With the use of this mobile application, it is aimed to increase the physical functions of the patients by reducing the level of anxiety and fear of movement.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were decided to undergo total knee replacement surgery with the diagnosis of osteoarthritis,
* Patients who will undergo elective surgery
* Patients who will undergo unilateral total knee replacement surgery for the first time
* Patients who can be communicated verbally
* Patients without any psychiatric disease
* Patients who use smartphones and agree to participate in the study

Exclusion Criteria:

* Patients under the age of 18
* Patients who have had previous total knee replacement surgery
* Patients who underwent total knee replacement with emergency surgery
* Patients who will undergo bilateral total knee replacement surgery
* Patients with a previous psychiatric diagnosis
* Patients with verbal communication disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-12-05 (Actual)

PRIMARY OUTCOMES:
State-Trait Anxiety Scale | 4 weeks
  The scale consists of two parts, a 20-item "state anxiety form" designed to determine what is felt at the moment, and a 20-item "trait anxiety form" designed to determine what is felt in general.
  It is a four-degree scale ranging from "Not at all" to "Totally". Scores range from 20 (low anxiety) to 80 (high anxiety).
Tampa Scale for Kinesiophobia | 4 weeks
  The scale consists of 17 items. The scale is a 4-point Likert type (1 = I strongly disagree, 4 = I completely agree) is used. The total score varies between 17-68. A high score on the scale indicates knesiophobia.
Knee injury and osteoarthritis outcome score-physical function short-form | 4 weeks
  The KOOS-PS scale consists of seven items. The items are intended to measure the degree of functionality of normal daily activities and more challenging activities. Each item scores between 0 "no difficulty" and 4 "very severe difficulty". The raw score is the sum of the scores given to these seven questions and ranges from 0 to 28. Higher scores indicate worse physical function.
Visual Analog Scale | 4 weeks
  The Visual Analog Scale is a widely used scale for the assessment of pain in patients. The patient marks his or her own pain on a 10 cm ruler with the words 'no pain' on one end and 'unbearable pain' on the other end.
Visual Analog Sleep Scale | 4 weeks
  This Visual Analog Sleep Scale measures the sleep quality of individuals. Each item in the scale is evaluated on a chart between 0 (left end) and 100 (right end) using the visual comparison technique. Scale scoring ranges from 0 to 1000. An increase in the score obtained from the scale indicates a decrease in sleep quality.
The Turkish Version of the Computer System Usability Questionnaire-Short Version | 4 weeks
  This questionnaire evaluates the usability of a software system with 13 items. Each item is scored as 1 (Strongly agree) - 7 (Strongly disagree).

CONTACTS AND LOCATIONS:
Overall Officials: Neziha Karabulut, PhD, Study Director — Ataturk University
Locations (1):
- Giresun University, Giresun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No